CLINICAL TRIAL: NCT00387595
Title: Family Atherosclerosis Counseling and Testing Project (FACT)
Brief Title: Family Atherosclerosis Counseling and Testing Project
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Jiri Frohlich, University of British Columbia
Other Study IDs: P02-0103
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: Family History; CAD; CAC; cIMT; CV Risk Factors
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Family history of early atherosclerotic disease in a first-degree relative [(FDR) sibling, parent or child] is an important risk factor for coronary artery and/or vascular disease. The risk increases ~ 2 - 7 times over that of general population. Increased thickness of the intima and media of carotid arterial wall, increased rate of plaque formation is an independent predictor of cardiovascular disease. Also it is shown that increased level of calcium deposition in the arterial wall is also associated with increased level of coronary artery narrowing. We will assess the occurrence and severity of abnormalities of intima media thickness (IMT) and/or plaque formation and increased calcium deposition in the coronary arteries and their relation to the well known traditional risk factors (plasma glucose, smoking, BMI, waist circumference, blood pressure, total cholesterol, low density lipoprotein, total cholesterol/high density lipoprotein ratio) and non-traditional risk factors (C-reactive protein, Lpa, homocysteine) in FDRs of index patients with early onset of heart or vascular disease and appropriate control population. Also to determine which of the above factor can assess IMT and Ca score better. This may help to reduce the cost of investigation, and to identify the population at high risk of developing cardiovascular disease, which may help the physicians to treat early on before cardiovascular complications occur. Also this may help to reduce the cost of invasive tests, hospital admissions and medical costs overall by reducing the morbidity and mortality.

DETAILED DESCRIPTION:
Objective: (i) To identify the differences between the "intervention" and "usual care" groups in Framingham risk scores, anthropometrical, biochemical parameters at baseline and at 24 months and compliance to prescribed regimens. Prevalence of maternal and paternal risk factors, DNA/mRNA profile and other risk factors may also be examined. (ii) To assess the relation between CIMT and psychosocial status with other conventional cardiovascular risk factors and serum levels of inflammatory markers in the "intervention" versus "usual care" groups over 2 years of follow up. (iii) Subjects that scored high on the emerging risk factors and IMT score will undergo CAC scanning. This will allow us to correlate the values of the CAC score in FDR's of patients with premature atherosclerosis to the IMT score and to the biochemical markers already captured in this study.

Method: (i) Index patients with premature atherosclerosis (angina with ECG changes, myocardial infarction, Coronary artery bypass grafting, Percutaneous transluminal coronary angioplasty, Peripheral vascular disease, Cerebro vascular disorders) in men below age 50yrs and women below age 60yrs at the time of the above mentioned adverse events will be identified from cardiac cath lab, healthy heart program St.Paul's and VGH, wards of St. Paul's hospital, heart function and transplant clinic and also from Cardiologists' offices, and will be asked to participate in the study. Those who volunteer to participate will be assessed for both the classical and emerging cardiovascular risk factors and asked for permission to approach their FDRs. The family of these index patients will be randomized using block randomization method (block of 4) in to usual care or intervention group. After recruitment of the patient, recruitment of their first degree relative will be undertaken. If present in the hospital during visiting hours, relatives will be approached in person by the study coordinator for participation in the study. Alternatively, relatives will be contacted by letter for participation, followed up by a telephone call.

FDRs and their spouses will undergo a comprehensive risk factor assessment including dietary, smoking, drinking and exercise habits. Data on past medical history, family history and treatment history will be collected. Anthropometric measurements (height, weight, waist circumference), blood pressure, heart rate and lipidemia markers will be recorded. Blood sample will be collected for biochemical measurements, which will include total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides, Apoprotein-B and A1, lipoprotein (a), homocysteine, C-reactive protein and glucose. Blood will be stored for future genetic analysis. Risk for future events will be estimated according to Framingham and or procam risk score. The same procedure will be repeated at the beginning and at the end of the 2-year period.

The participants will be divided into "intervention" and "usual care" groups. The intervention group will receive a risk assessment summary, with a copy to their family physician. Recommendations for treatment of modifiable risk factors to targets (blood pressure control, lipids, glucose, and smoking cessation) and counseling will be carried out. Regular follow up of study participants at 3 and 6 months will be made and patient will be called over phone at 4 and 8 months for lifestyle counseling and all participants will be reassessed at 2 year. The usual care group will receive an initial risk assessment summary along with their diet, exercise and other risk assessments using the questionnaire. The risk assessment summary will be mailed to the patient and to their family physicians with a note highlighting the abnormal results and will be asked to discuss this with them. The same procedure will be repeated at the end of the 2-year period. The comparison of intervention and usual care groups will be made at 24 months after their initial assessment for their health and risk factor profile.

(ii) Those participants older than 30 yrs with >10% risk score who volunteer to participate in FACT phase 2 study will be asked to sign a consent for the IMT study and be given the psychosocial questionnaire to complete and asked to bring it back at the time of their IMT visit. IMT will be measured by experienced technicians using HP Pointrex ultrasound scanner. This takes about 45 minutes. The data will be analysed by the experienced sonographer and stored offline for future use. A second scan will be performed two years later.

(iii) Subjects already enrolled in the study that underwent IMT scan for the baseline visit will be selected as candidates for this procedure. Patients who meet the above criteria will be selected form both the "intervention" and "usual care" group; contacted by mail/phone and asked to participate in this portion of the study. If, they agree, patients will be given a new consent form to sign and after the consenting is done, an appointment for the CAC scan is made.

The subject will be asked to abstain from caffeine or caffeine-containing products the day of the scan in order to ensure an optimal rest heart beat < 80bpm. No other preparation is necessary for this procedure. The total length of this appointment is about 30 minutes, and most of this time is required to place ECG patches and to properly position the subject. The actual scan takes only 20 seconds. The technician will ask the patient to hold his breath for approximately 20 seconds while the scan is performed. The CAC scan will be administered by a trained technician at the Canada Diagnostic Centre located at 136-55 West 12th Avenue in Vancouver, BC. Except for the small amount of radiation the patient will be exposed to during this procedure there are no other known risks associated with this scan.

ELIGIBILITY:
Inclusion Criteria:

* First degree relatives of patients with early onset of cardiovascular disease (men<50 and women<60 years of age).

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Frohlich, Principal Investigator — University of British Columbia

REFERENCES:
- [Derived] Taraboanta C, Hague CJ, Mancini GB, Forster BB, Frohlich J. Coronary artery calcium findings in asymptomatic subjects with family history of premature coronary artery disease. BMC Cardiovasc Disord. 2012 Jul 17;12:53. doi: 10.1186/1471-2261-12-53. PMID 22805651